CLINICAL TRIAL: NCT00230230
Title: SCH 486757 vs Codeine and Placebo in Subjects With Persistent Postviral Cough
Brief Title: Comparison of SCH 486757 to Codeine and Placebo in Subjects With Persistent Postviral Cough (Study P03069AM2)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03069
Record Dates: First submitted 2005-09-22; First posted 2005-09-30 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — 8-(bis(2-chlorophenyl)methyl)-3-(2-pyrimidinyl)-8-azabicyclo(3.2.1)octan-3-ol

INTERVENTIONS:
Drug: SCH 486757

SUMMARY:
This randomized, multicenter, parallel-group, double-blind, double-dummy, placebo- and active-controlled study will evaluate the efficacy and safety of SCH 486757 in subjects with persistent cough resulting from a recent viral upper respiratory infection (URI). The primary objective is to assess the efficacy of SCH 486757 administered at a dose of 100 mg twice daily for 5 days in the reduction of cough severity score compared with placebo. The key secondary objective is to evaluate the reduction in the number of coughs with SCH 486757 compared with placebo. Because codeine is a widely used as a cough medication, it is included as a treatment arm in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to <65 years of age, of either sex, and of any race.
* At the prescreening visit (Visit 1), subjects must have a history of a persistent cough resulting from a recent viral URI.
* Subjects must be sufficiently clinically symptomatic at the screening visit (Visit 2).
* At the Baseline/Treatment Day 1 Visit (Visit 3), subjects must demonstrate an average cough severity score of at least 2 (moderate).
* Subjects must be in good health, free of any clinically significant disease, other than cough, that might interfere with the study schedule, evaluation, or interpretation of study-derived data.
* Subjects must be willing to give written informed consent and able to adhere to dose and visit schedules.
* Clinical laboratory tests (complete blood count, blood chemistries, and urinalysis) and electrocardiograms must be within normal limits or clinically acceptable to the investigator.
* Female subjects of childbearing potential must be using a medically accepted method of birth control.
* Female subjects of childbearing potential must have a negative serum pregnancy test (beta-hCG) (prescreening sample).

Exclusion Criteria:

* Subjects who are pregnant or nursing females.
* Subjects with a history of hypersensitivity to the study medications or to their excipients.
* Subjects who have used any study medication, including placebo, in an investigational protocol within 30 days prior to the prescreening visit (Visit 1).
* Subjects receiving concurrent prohibited medications, unless they observe the washout period prior to the screening and baseline visits (Visits 2 and 3).
* Subjects who are family members of the investigational study staff involved with this study.
* Subjects previously enrolled into this study (ie, signed informed consent).
* Subjects with current evidence of clinically significant pulmonary (especially conditions that involve coughing), hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune, or other disease that precludes the subject's participation in the study. In particular, diabetics, uncontrolled hypertensives, and subjects with clinically significant cardiomyopathy, prostatic hypertrophy, glaucoma, and psychiatric disorders are to be excluded from participation in this study. Particular attention should be given to exclude subjects with conditions that would currently interfere with the absorption, distribution, metabolism, or excretion of the study medication or interfere with the subject's ability to reliably complete the diary card.
* Subjects with asthma or chronic obstructive pulmonary disease who require chronic use of inhaled or systemic corticosteroids.
* Subjects with current or history of frequent clinically significant sinusitis or chronic purulent postnasal drip.
* Subjects with a history of allergies to more than two classes of medications.
* Subjects whose ability, in the opinion of the investigator or designee, to provide informed consent is compromised.
* Subjects with a history of noncompliance with medications or treatment protocols, or with a history of drug abuse.
* Current smokers, ex-smokers who stopped smoking in the previous 6 months, or subjects with a cumulative smoking history >10 pack-years will be excluded. (Pack-years is a way to measure the amount a person has smoked over a long period of time. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked, eg, a 10 pack-year history is equal to smoking 1 pack per day for 10 years or 2 packs per day for 5 years, etc.)
* Subjects with current reflux disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2005-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

REFERENCES:
- [Result] Woodcock A, McLeod RL, Sadeh J, Smith JA. The efficacy of a NOP1 agonist (SCH486757) in subacute cough. Lung. 2010 Jan;188 Suppl 1:S47-52. doi: 10.1007/s00408-009-9197-8. PMID 19937046